CLINICAL TRIAL: NCT01843036
Title: Second RCT Evaluation of the Durham Connects Universal Newborn Nurse Home Visiting Program
Brief Title: Durham Connects RCT Evaluation II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Duke Endowment (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Coalition for Evidence-Based Policy (Unknown); Laura and John Arnold Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00052735; Pro00017478 (Other: Duke University Medical System IRB); 1R01HD069981 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Unspecified Child Maltreatment, Suspected; Unspecified Child Maltreatment, Confirmed
Keywords: Child Abuse; Child Neglect; Child Emergency Medical Care Presentations; Child Well-Care Compliance; Mother Well-Care Compliance; Mother Emergency Medical Care Presentations; Mother Mental Health; Family Connections to Community Resources; Parent-Child Relationship Quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durham Connects Eligible (Experimental): From January 1, 2014 - June 30, 2014, all odd-birth-date residential births in Durham County, North Carolina will be randomly assigned to receive the Durham Connects nurse home visiting program.
  Interventions: Other: Durham Connects
- Control (No Intervention): From January 1, 2014 - June 30, 2014, all even-birth-date residential births in Durham County, North Carolina will be randomly assigned to a control group condition. These families will be assigned to receive services as usual and serve as the randomized comparison group for evaluating Durham Connects program impact.

INTERVENTIONS:
Other: Durham Connects — Durham Connects begins with a visit during the birthing hospital stay, followed by 1-3 nurse home visits between 4-12 weeks of infant age, and then a follow-up contact one month later. During the visits, the nurse engages with the mother and completes a health and psychosocial assessment, during which she systematically assesses risk and family needs in 12 important empirically-derived areas of family functioning across 4 domains (i.e. - healthcare, parenting/childcare, family violence/safety, and maternal well-being). For each domain found to be at risk, the nurse intervenes directly to support the mother (mild risk) or connects the mother with matched community resources as needed to address individualized long-term family needs (moderate or severe risk).
  Arms: Durham Connects Eligible

SUMMARY:
The aim of this randomized controlled trial (RCT) is to conduct a second, independent evaluation the implementation and impact of the Durham Connects (DC) brief universal nurse home-visiting program to prevent child maltreatment and improve child and family health and well-being. Durham Connects is the first home-visiting program that is designed to prevent child maltreatment and improve health and well-being outcomes in an entire community population.

Program evaluation will test four hypotheses: 1) The program can be implemented with population reach, fidelity to the manualized intervention protocol, and reliability in assessment of family risk; 2) Random assignment to the Durham Connects program will be associated with lower rates of child maltreatment and emergency department maltreatment-related injuries, better pediatric care, better parental functioning, and better child well-being than assignment as control; 2) Intervention effect sizes will be larger for higher-risk groups; and 3) Community resource use and enhanced family functioning will mediate the positive impact of Durham Connects on outcomes.

DETAILED DESCRIPTION:
The Durham Connects program is an innovative, community-based, universal nurse home-visiting program that aims to lower the population rate of child maltreatment and improve child and family health and well-being. The Durham Connects Program is implemented jointly by the Durham County (North Carolina) Health Department, the Center for Child & Family Health, and Duke University. It is designed to be brief and inexpensive per family so that communities can afford its costs. Its goals are consistent with those of more intensive nurse home-visiting programs: 1) to connect with the mother in order to enhance maternal skills and self-efficacy; and 2) to connect the mother with needed community services such as health care, child care, mental health care, and financial and social support; so that 3) the mother can connect with her child.

DC achieves population reach by engaging all families within the community, rapidly triaging families based on identified risk to concentrate resources to families with greater needs, and connecting those families with significant nurse-identified risk to matched community programs and services to provide long-term support and a first step into the community system of care. The program consists of 4-7 manualized intervention contacts, including 1) a hospital birthing visit when a staff member communicates the importance of community support for parenting and schedules an initial home visit; 2) 1-3 nurse home visits between 3-12 weeks of infant age to provide physical assessments for infant and mother, intervention and education, assessment of family-specific needs, and for families with significant nurse-identified risk, connections to matched community resources to provide longer-term support; 3) 1-2 nurse contacts with community service providers to facilitate successful connections; and 4) a telephone follow-up one month after case closure to review consumer satisfaction and community connection outcomes. With family consent, letters from the program reporting on the visit are also provided to also connect families to maternal and infant healthcare providers for ongoing support.

During home visits, the nurse engages the mother (and father, when possible) to provide brief educational interventions for all families (e.g., safe sleep) and utilizes a high-inference approach to assess family needs across 12 empirically-derived factors linked to child health and well-being: Healthcare: parent health, infant health, health care plans; Parenting/childcare: childcare plans, parent-infant relationship, management of infant crying; Family violence/safety: material supports, family violence, maltreatment history; and Parent well-being: depression/anxiety, substance abuse, social/emotional support.

The nurse scores each of the 12 factors and intervenes accordingly. A score of 1 (low risk) receives no subsequent intervention. A score of 2 (moderate risk) receives short-term, nurse-delivered intervention over 1-2 sessions. For a score of 3 (high risk) the nurse connects the family to matched community resources tailored to address that particular risk (such as, treatment for postpartum depression, a DSS social worker exclusively serving Durham Connects families for enrollment in Medicaid or food stamps, a multi-year home visiting program for long-term parent support). The nurse also provides follow up to make sure that each connection "sticks," requiring additional contacts with the family or community agency. A score of 4 (imminent risk) receives emergency intervention (<1% of cases). A final contact four weeks after case closure ascertains community connection outcomes and whether further problem solving is needed to address new or existing needs.

From January 1, 2014, through June 30, 2014, all residential births in Durham County, North Carolina (~1600) will randomly assigned according to birthdate, with odd-birth-dates assigned to receive DC. Even-birth-dates will be assigned to receive services-as-usual and serve as the randomized control group. All eligible families (i.e., families living in Durham County giving birth at one of the two county hospitals) were included with experimental rigor, and without exception, but with ethical care for confidentiality. Hospital discharge records were utilized to confirm eligibility for all RCT families. Program implementation will be evaluated for all odd-birth-date families. The Duke University Health System Institutional Review Board approved all RCT implementation and evaluation procedures.

Completely independent of program implementation, all RCT families were contacted and invited to participate in an independent evaluation of DC short-term impact at infant age 6 months (interviews completed between infant ages 6-8 months). Eligible RCT families were identified using short-form public birth records (i.e., resident Durham County births at one of the two county birthing hospitals) without consideration for intervention participation or adherence. RCT families were contacted and invited to participate in a descriptive research study about family community service use and child development. Families were blind to study goals, and home interviewers were blind to family DC participation status.

ELIGIBILITY:
Inclusion Criteria:

* Infant born between January 1, 2014 and June 30, 2014
* Infant born at a Durham County, North Carolina (NC) hospital (Duke or Durham Regional)
* Family of infant resides in Durham County, NC

Exclusion Criteria:

* Infant born before January 1, 2014 or after June 30, 2014
* Infant not born at a Durham County, NC hospital (Duke or Durham Regional)
* Family of infant resides outside of Durham County, NC

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1650 (Estimated)
Dates: Start 2014-01; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
DSS Investigated and Substantiated Child Maltreatment Rates | 0 - 12 Years of Child Age
  North Carolina Department of Social Services (DSS) reported lifetime cases of investigated and substantiated maltreatment caseness

SECONDARY OUTCOMES:
Child Emergency Room (ER) Presentation Rates | 0 - 12 Years of Child Age
  Lifetime child emergency department visits reported in hospital administrative records.
Child Overnight Stays in Hospital | 0 - 12 Years of Child Age
  Lifetime child overnight stays in hospital for all overnight stays unrelated to the birthing stay reported in hospital administrative records.
Mother Postnatal Well-Care Compliance Rates | 0-6 Months Postnatal
  Rates of mother compliance with postnatal well-care as reported by the mother
Child Postnatal Well-Care Compliance Rates | 0-6 Months Postnatal
  Rates of infant compliance with postnatal well-care health checks as reported by the mother
Mother Emergency Room (ER) Presentation Rates | 0 - 12 Years of Child Age
  Total mother emergency department visits as reported in hospital administrative records.
Mother Overnight Stays in Hospital | 0 - 12 Years of Child Age
  Total mother overnight stays in hospital for all overnight stays unrelated to the birthing stay reported in hospital administrative records.
Mother Mental Health | 0-6 Months Postnatal
  Rates of mother depressive symptoms and anxiety symptoms as reported by the mother
Family Connections to Community Services/Resources | 0-6 Months Postnatal
  Rates of family connections to community resources and services as reported by the mother
Mother Parenting Behaviors | 0-6 Months Postnatal
  Rates of mother positive and negative parenting behaviors as reported by the mother

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Dodge, Ph.D., Principal Investigator — Duke University; Robert Murphy, Ph.D., Principal Investigator — Center for Child & Family Health; Karen O'Donnell, Ph.D., Principal Investigator — Center for Child & Family Health; W. Benjamin Goodman, Ph.D., Principal Investigator — Duke University
Locations (1):
- Center for Child and Family Policy, Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodge KA, Goodman WB, Bai Y, Best DL, Rehder P, Hill S. Impact of a universal perinatal home-visiting program on reduction in race disparities in maternal and child health: Two randomised controlled trials and a field quasi-experiment. Lancet Reg Health Am. 2022 Aug 23;15:100356. doi: 10.1016/j.lana.2022.100356. eCollection 2022 Nov. PMID 36778074
- [Result] Dodge KA, Goodman WB, Bai Y, O'Donnell K, Murphy RA. Effect of a Community Agency-Administered Nurse Home Visitation Program on Program Use and Maternal and Infant Health Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914522. doi: 10.1001/jamanetworkopen.2019.14522. PMID 31675088
- See also: Family Connects International Website — http://familyconnects.org/
- See also: Center for Child and Family Policy, Duke University — http://childandfamilypolicy.duke.edu/
- See also: Center for Child & Family Health — http://www.ccfhnc.org/